CLINICAL TRIAL: NCT04213612
Title: Phase I Study of Pegylated Liposomal Doxorubicin Combined With Cyclophosphamide and Vincristine in Treatment Progress, Relapse, and Refractory Solid Tumors in Children
Brief Title: DCV in the Treatment of Recurrence and Refractory Childhood Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-1-19
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Unrecognized Condition
MeSH Terms: interventions — liposomal doxorubicin; Cyclophosphamide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLD+CTX+VCR (Experimental): CTX 1g/m2/d，D1-2 VCR 1.5mg/m2，D1
  Interventions: Drug: pegylated liposomal doxorubicin, cyclophosphamide, vincristine,

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin, cyclophosphamide, vincristine, — PLD 40mg/m2 ; PLD 50mg/m2 ; PLD 60mg/m2 ; Maximum tolerated dose； Dose-limiting toxicity
  Other Names: Doxorubicin Hydrochloride Liposome Injection

SUMMARY:
Doxorubicin is an anthracycline antibiotic that is part of the standard treatment for many pediatric malignancies, but its long-term cardiotoxicity cannot be ignored. Without affecting overall survival, in order to improve the quality of life of childhood tumor survivors and reduce cardiotoxicity, drugs with less cardiotoxicity should be selected; compared with ordinary doxorubicin, PEGylated doxorubicin (PLD ) The biggest advantage is the low cardiotoxicity.

PEGylated doxorubicin (Caelyx®) has undergone a Phase I dose climbing clinical trial in children with solid tumors. The drug is safe by testing PK. The results of Phase II clinical studies of Caelyx® in children with progressive soft tissue sarcoma show that the drug is safe. Domestically produced PEGylated doxorubicin has no data on childhood tumors in China. Therefore, we plan to conduct a phase I study in pediatric solid tumors of pegylated doxorubicin combined with cyclophosphamide, vincristine, relapsed, and refractory childhood solid tumors. Maximum tolerated dose and effectiveness of stellate in children with solid tumors, thus laying the foundation for future phase II / III clinical studies

DETAILED DESCRIPTION:
Purpose of Phase I:

the main purpose: To evaluate the safety of PLD in combination with cyclophosphamide, vincristine, regenerative, and refractory solid tumors in children, including dose absorption toxicity (DLT)

Secondary purpose:

* determine the appropriate maximum tolerated dose (MTD) and /or PLD for further clinical studies in this patient population;
* Describe the antitumor activity of PLD combined with cyclophosphamide and vincristine in children with advanced solid tumors or primary CNS tumors;

Exploratory purpose:

Effectiveness of PLD combined with cyclophosphamide and vincristine in treatment progress, relapse, and refractory solid tumors in children.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 1-18 years;
* 2) ECOG PS score: 0-1 points;
* 3) Patients with solid tumors confirmed by histopathology in children;
* 4) Patients who have progressed, relapsed, or are refractory after first-line treatment (there is no complete or partial response after recent treatment);
* 5) Must have at least one measurable lesion as defined by the RECIST standard;
* 6) Expected survival time ≥ 6 months;
* 7) Heart function:

  1. Cardiac ultrasound detection LVEF ≥ 50%;
  2. EKG indicates no myocardial ischemia;
  3. no history of arrhythmia requiring drug intervention before enrollment;
* 8) Patients must fully recover from the acute toxic effects of all previous anti-cancer chemotherapy:

  1. Myelosuppressive chemotherapy: at least 21 days after the last myelosuppressive chemotherapy (42 days if nitrosourea was used earlier);
  2. Experimental drugs or anti-cancer therapies other than chemotherapy: Do not use within the first 28 days of the planned start of doxycycline. Full recovery from the clinically significant toxicity of the therapy must be clearly identified;
  3. Hematopoietic growth factor: at least 14 days after the last dose of long-acting growth factor or 3 days after the last dose of short-acting growth factor;
  4. immunotherapy: at least 42 days after completing any type of immunotherapy (except steroids), such as immune checkpoint inhibitors and tumor vaccines;
  5. X-ray therapy (XRT): at least 14 days after local palliative XRT ( small range of mouth); if other solid bone marrow (BM) irradiation, including prior radioactive iodized meta-iodobenzidine (131I-MIBG) treatment, You must end at least 42 days;
  6. Stem cell infusion without total body irradiation (TBI): There is no evidence of active graft-versus-host disease, and transplantation or stem cell infusion must end at least 56 days;
* 9) For patients who are not known to have BM:

  1. Absolute neutrophil count (ANC) ≥ 1.0 × 109 / L;
  2. Platelet count ≥100.0 × 109 / L;
  3. hemoglobin ≥90 g / L;
* 10) Liver and kidney function should meet the following standards:

  1. Bilirubin (combined + unbound total) ≤ 2.5 × upper limit of normal value (ULN) (corresponding to age), patients with Gilbert's syndrome can be enrolled according to the researchers' judgment
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN;
  3. Estimated glomerular filtration rate ≥ 30 mL / min / 1.73 m2 or serum creatinine (Cr) ≤ 1.5ULN;
* 11) During the participation in the study, be able to comply with outpatient treatment, laboratory monitoring and necessary clinical visits;
* 12) The parent/ guardian of the child or adolescent subject has the ability to understand, agree, and sign the research informed consent (ICF) and applicable child consent form before initiating any protocol-related procedures; subject to parent/ guardian consent Candidates have the ability to express consent (if applicable).

Exclusion Criteria:

* 1) Previous or concurrent active clinical cardiovascular disease including congenital heart disease or pericardial disease, history of heart failure, myocardial infarction, coronary heart disease, heart valve disease, cardiomyopathy, arrhythmia (including persistent atrial fibrillation, Complete left bundle branch block, frequent ventricular early); or the QT interval (QTc) after the current corrected heart rate is extended> 480 milliseconds;
* 2) previous severe skin diseases;
* 3) previous allergic asthma or severe allergic disease;
* 4) Poorly controlled hypertension and diabetes;
* 5) Have a history of other tumors, except for cured cervical cancer or skin basal cell carcinoma;
* 6) Patients with hepatitis B surface antigen-positive;
* 7) Patients infected with HIV or syphilis;
* 8) Patients who have received organ transplants in the past;
* 9) Uncontrolled active systemic bacterial, viral or fungal infections;
* 10) Contraindications to high-dose hormone use, such as uncontrollable high blood sugar, gastric ulcer or mental illness;
* 11) Patients who have used a total cumulative dose of doxorubicin ≥ 450 mg / m2, or a total cumulative dose of epirubicin ≥ 550 mg / m2, or previously used anthracyclines to cause heart disease;
* 12) Have a serious neurological or psychiatric history, including epilepsy or autism.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-12-30 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | At the end of Cycle 1 (each cycle is 21 days)
  Maximum tolerated dose

SECONDARY OUTCOMES:
Adverse event | through study completion, an average of 1 year
  Hematological and non-hematological toxicity (NCI CTCAE v5.0)
Objective Response Rate | At the end of Cycle 2 (each cycle is 21 days)
  Complete remission + partial remission

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University CancerCenter

REFERENCES:
- [Background] Singal PK, Deally CM, Weinberg LE. Subcellular effects of adriamycin in the heart: a concise review. J Mol Cell Cardiol. 1987 Aug;19(8):817-28. doi: 10.1016/s0022-2828(87)80392-9. No abstract available. PMID 3320376
- [Background] Von Hoff DD, Layard MW, Basa P, Davis HL Jr, Von Hoff AL, Rozencweig M, Muggia FM. Risk factors for doxorubicin-induced congestive heart failure. Ann Intern Med. 1979 Nov;91(5):710-7. doi: 10.7326/0003-4819-91-5-710. PMID 496103
- [Background] Swain SM, Whaley FS, Ewer MS. Congestive heart failure in patients treated with doxorubicin: a retrospective analysis of three trials. Cancer. 2003 Jun 1;97(11):2869-79. doi: 10.1002/cncr.11407. PMID 12767102
- [Background] Abu Lila AS, Ishida T, Kiwada H. Recent advances in tumor vasculature targeting using liposomal drug delivery systems. Expert Opin Drug Deliv. 2009 Dec;6(12):1297-309. doi: 10.1517/17425240903289928. PMID 19780711
- [Background] Gabizon AA. Selective tumor localization and improved therapeutic index of anthracyclines encapsulated in long-circulating liposomes. Cancer Res. 1992 Feb 15;52(4):891-6. PMID 1737351
- [Background] Northfelt DW, Martin FJ, Working P, Volberding PA, Russell J, Newman M, Amantea MA, Kaplan LD. Doxorubicin encapsulated in liposomes containing surface-bound polyethylene glycol: pharmacokinetics, tumor localization, and safety in patients with AIDS-related Kaposi's sarcoma. J Clin Pharmacol. 1996 Jan;36(1):55-63. doi: 10.1002/j.1552-4604.1996.tb04152.x. PMID 8932544
- [Background] O'Brien ME, Wigler N, Inbar M, Rosso R, Grischke E, Santoro A, Catane R, Kieback DG, Tomczak P, Ackland SP, Orlandi F, Mellars L, Alland L, Tendler C; CAELYX Breast Cancer Study Group. Reduced cardiotoxicity and comparable efficacy in a phase III trial of pegylated liposomal doxorubicin HCl (CAELYX/Doxil) versus conventional doxorubicin for first-line treatment of metastatic breast cancer. Ann Oncol. 2004 Mar;15(3):440-9. doi: 10.1093/annonc/mdh097. PMID 14998846
- [Background] Schmitt CJ, Dietrich S, Ho AD, Witzens-Harig M. Replacement of conventional doxorubicin by pegylated liposomal doxorubicin is a safe and effective alternative in the treatment of non-Hodgkin's lymphoma patients with cardiac risk factors. Ann Hematol. 2012 Mar;91(3):391-7. doi: 10.1007/s00277-011-1308-y. Epub 2011 Aug 18. PMID 21850390
- [Background] Judson I, Radford JA, Harris M, Blay JY, van Hoesel Q, le Cesne A, van Oosterom AT, Clemons MJ, Kamby C, Hermans C, Whittaker J, Donato di Paola E, Verweij J, Nielsen S. Randomised phase II trial of pegylated liposomal doxorubicin (DOXIL/CAELYX) versus doxorubicin in the treatment of advanced or metastatic soft tissue sarcoma: a study by the EORTC Soft Tissue and Bone Sarcoma Group. Eur J Cancer. 2001 May;37(7):870-7. doi: 10.1016/s0959-8049(01)00050-8. PMID 11313175
- [Background] Beverdam A, Meijlink F. Expression patterns of group-I aristaless-related genes during craniofacial and limb development. Mech Dev. 2001 Sep;107(1-2):163-7. doi: 10.1016/s0925-4773(01)00450-6. PMID 11520673
- [Background] Wagner HE, Gilg M, Baer HU. [Characteristics of tumor diseases in patients with colorectal cancer]. Helv Chir Acta. 1993 Mar;59(4):701-3. German. PMID 8473195
- [Derived] Lu S, Wang J, Huang J, Sun F, Zhu J, Que Y, Li H, Guo Y, Cai R, Zhen Z, Sun X, Zhang Y. Pegylated liposomal doxorubicin combined with cyclophosphamide and vincristine in pediatric patients with relapsed/refractory solid tumor: a single-arm, open-label, phase I study. EClinicalMedicine. 2024 Jun 20;73:102701. doi: 10.1016/j.eclinm.2024.102701. eCollection 2024 Jul. PMID 39007065
- See also: Singal, P.K., C.M. Deally and L.E. Weinberg, Subcellular effects of adriamycin in the heart: a concise review. J Mol Cell Cardiol, 1987. 19(8): p. 817-28. — http://www.ncbi.nlm.nih.gov/pubmed/3320376
- See also: Von Hoff, D.D., et al., Risk factors for doxorubicin-induced congestive heart failure. Ann Intern Med, 1979. 91(5): p. 710-7 — https://www.ncbi.nlm.nih.gov/pubmed/496103
- See also: Swain, S.M., F.S. Whaley and M.S. Ewer, Congestive heart failure in patients treated with doxorubicin: a retrospective analysis of three trials. Cancer, 2003. 97(11): p. 2869-79 — https://www.ncbi.nlm.nih.gov/pubmed/12767102
- See also: Abu A L, Ishida T, Kiwada H. Recent advances in tumor vasculature targeting using liposomal drug delivery systems.[J]. Expert Opinion on Drug Delivery, 2009, 6(12):1297. — https://www.ncbi.nlm.nih.gov/pubmed/19780711
- See also: Gabizon AA. Selective tumor localization and improved therapeutic index of anthracyclines encapsulated in long-circulating liposomes[J]. Cancer Research, 1992, 52(4):891-896. — https://www.ncbi.nlm.nih.gov/pubmed/1737351
- See also: Northfelt D W, Martin F J, Working P, et al. Doxorubicin Encapsulated in Liposomes Containing Surface-Bound Polyethylene Glycol: Pharmacokinetics, Tumor Localization, and Safety in Patients — https://www.ncbi.nlm.nih.gov/pubmed/8932544
- See also: Reduced cardiotoxicity and comparable efficacy in a phase III trial of pegylated liposomal doxorubicin HCl (CAELYX/Doxil) versus conventional doxorubicin for first-line treatment of metastatic breast cancer. — https://www.ncbi.nlm.nih.gov/pubmed/14998846
- See also: Schmitt, C.J., et al., Replacement of conventional doxorubicin by pegylated liposomal doxorubicin is a safe and effective alternative in the treatment of non-Hodgkin's lymphoma patients with cardiac risk factors. Ann Hematol, 2012. 91(3): p. 391-7 — https://www.ncbi.nlm.nih.gov/pubmed/21850390
- See also: Randomised phase II trial of pegylated liposomal doxorubicin (DOXIL/CAELYX) versus doxorubicin in the treatment of advanced or metastatic soft tissue sarcoma: a study by the EORTC Soft Tissue and Bone Sarcoma Group — https://www.ncbi.nlm.nih.gov/pubmed/11313175
- See also: Marina, N.M., et al., Dose escalation and pharmacokinetics of pegylated liposomal doxorubicin (Doxil) in children with solid tumors: a pediatric oncology group study. Clin Cancer Res, 2002. 8(2): p. 413-8. — https://www.researchgate.net/publication/11520673_Marina_NM_Cochrane_D_Harney_E_Zomorodi_K_Blaney_S_Winick_N_Bernstein_M_Link_MPDose_escalation_and_pharmacokinetics_of_pegylated_liposomal_doxorubicin_Doxil_in_children_with_solid_tumors_a_Pediatric_On
- See also: Munoz, A., et al., Pegylated liposomal doxorubicin hydrochloride (PLD) for advanced sarcomas in children: preliminary results. Pediatr Blood Cancer, 2004. 43(2): p. 152-5. — https://www.researchgate.net/publication/8473195_Pegylated_liposomal_doxorubicin_hydrochloride_PLD_for_advanced_sarcomas_in_children_Preliminary_results